CLINICAL TRIAL: NCT05514015
Title: A Prospective, Randomized, Multicenter Clinical Trial Comparing the Efficacy and Safety of Rituximab Combined With Corticosteroids or Rituximab Monotherapy in Primary Membranous Nephropathy
Brief Title: Clinical Study of Rituximab Combined With Corticosteroids or Rituximab Monotherapy in the Treatment of Primary Membranous Nephropathy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wei Chen, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLK-202302
Record Dates: First submitted 2022-08-14; First posted 2022-08-24 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Primary Membranous Nephropathy
Keywords: rituximab; Primary membranous nephropathy; rituximab combined with corticosteroids; safety; remission
MeSH Terms: interventions — Adrenal Cortex Hormones; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): rituximab combined with corticosteroids treatment group
  Interventions: Drug: rituximab combined with corticosteroids
- Control arm (Active Comparator): Rituximab monotherapy treatment
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab combined with corticosteroids — Induction therapy:
  Rituximab intravenous infusion of 1g, d1, d15, combined with glucocorticoid therapy, oral prednisolone, initial dose of 0.5mg/(kg·d), once a day, after 8 weeks of treatment, reduce by 5mg every 4 weeks until 0.25mg/kg, this dose was maintained for 8 weeks, and then reduced by 2.5mg every 4 weeks, until 5-10mg is maintained, and the total course of treatment was about one year or so;
  Other Names: Intervention arm
  Arms: Intervention arm
Drug: rituximab — Control group (treated with Rituximab monotherapy treatment) :Rituximab intravenous infusion of 1g, d1, d15
  Other Names: Control arm
  Arms: Control arm

SUMMARY:
This was a prospective, randomized, multicenter clinical trial. Seventy-eight patients with primary membranous nephropathy (PMN) were randomly divided into intervention or control group. Intervention group was given rituximab combined with corticosteroids in induction therapy and the control group was given rituximab monotherapy. After 6 months, patients who had decreased 24h urinary protein by > 25% but did not achieve CR were given rituximab maintenance therapy. The complete response rate at 12 months was measured.

DETAILED DESCRIPTION:
Study design A prospective, randomized , multicenter clinical study

Outcomes

* Primary objective To evaluate the efficacy of rituximab combined with corticosteroids or rituximab monotherapy in primary membranous nephropathy
* Secondary Objectives The safety of rituximab combined with corticosteroids or rituximab monotherapy in primary membranous nephropathy;

Primary outcome The complete response rate at 12 months;

* Secondary outcomes

  1. Response rates at 6, 12, 18 and 24 months (including the proportion of participants with complete response and partial response);
  2. Median remission time;
  3. Proportion of patients without recurrence at 12, 18 and 24 months;
  4. Median non-recurrence time;
  5. Cumulative dose of glucocorticoids;
  6. CD19+ cell count, anti-PLA2R antibody expression level;
  7. Renal function index: eGFR;
  8. Incidence of adverse events;

     Study population Seventy-eight male or female treatment-naïve primary membranous nephropathy (PMN) patients

     Description of the study intervention Intervention group: rituximab combined with corticosteroids: 39 cases. Patients are pretreated with diphenhydramine and dexamethasone 30-60 minutes before rituximab infusion.
* Induction therapy:

Rituximab intravenous infusion of 1g, d1, d15, combined with glucocorticoid therapy, oral prednisolone, initial dose of 0.5mg/(kg·d), once a day, after 8 weeks of treatment, reduce by 5mg every 4 weeks until 0.25mg/kg, this dose was maintained for 8 weeks, and then reduced by 2.5mg every 4 weeks, until 5-10mg is maintained, and the total course of treatment was about one year or so;

- Consolidation therapy after 6 months: Patients who achieve CR do not require consolidation therapy; Patients who had a 24-hour reduction in proteinuria >25% but did not achieve CR received an additional course of rituximab 1g, D1, D15 (independent of CD19+ cell count).

Patients with less than 25% decrease in proteinuria in 24 hours do not require continued medical therapy, and were considered as treatment failure and withdraw from the trial.

Control group: Rituximab monotherapy: 39 cases,

- Treatment regimen: 30-60 minutes before intravenous infusion of rituximab, diphenhydramine 20mg intramuscularly and dexamethasone 5mg intravenously were given for pretreatment.

* Induction therapy:Rituximab intravenous infusion of 1g, d1, d15
* Consolidation therapy after 6 months:

Patients who achieve CR do not require consolidation therapy; Patients who had a 24-hour reduction in proteinuria >25% but did not achieve CR received an additional course of rituximab 1g, D1, D15 (independent of CD19+ cell count).

Patients with less than 25% decrease in proteinuria in 24 hours do not require continued medical therapy, and were considered as treatment failure and withdraw from the trial.

The duration of the entire clinical study was 36 months from the date of project initiation.

Duration of visits: 2 years

ELIGIBILITY:
Inclusion Criteria

1. Men and women aged 18-75 years;
2. Patients diagnosed as primary membranous nephropathy (PMN) by renal biopsy;
3. After treatment with ACE inhibitors or ARBs for at least 3 months, the following two points were met (unless intolerance to ACE inhibitors or ARBs, contraindications, hypotension that may cause side effects, or the investigator judged that the patient was not suitable for RAS inhibitors):

(1) Those who have an average 24-hour urine protein ≥ 3.5g twice a week, or an average 24-hour urine protein ≥ 5g twice in 14 days, the requirement of RASi for at least 3 months is not required (2) Blood pressure≤ 130/80mmHg, 4. Glomerular filtration rate (eGFR) ≥30mL/min/1.73m2 (calculated according to the CKD-EPI formula) 5. If female, must be postmenopausal or postoperatively infertile or on medical contraception (considering the potential risk of thromboembolism in patients with kidney disease); 6. Subjects voluntarily signed the informed consent form;

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus or type 2 diabetes mellitus complicated with diabetic nephropathy. Patients with a recent history of steroid-induced diabetes were eligible if renal biopsies show no evidence of secondary diabetic nephropathy within 6 months before the screening period
2. Patients with secondary membranous nephropathy (such as hepatitis B and C, systemic lupus erythematosus, drug therapy, malignant tumors and other secondary causes);
3. Previous treatment with rituximab, steroids, alkylating agents, calcineurin inhibitors, synthetic ACTH, mycophenolate (MMF), and azathioprine;
4. Receipt of any other study medication (within the last month);
5. Suspected or known allergy or immune reaction to rituximab, corticosteroids or any of their components (including excipients);
6. Active infection, such as active hepatitis B or hepatitis C, tuberculosis (evidence of active tuberculosis infection within 1 year), or human immunodeficiency virus HIV infection (positive for anti-HIV antibodies), etc.
7. A history of immunodeficiency, including other acquired or congenital immunodeficiency diseases, or organ transplantation;
8. Females with a positive pregnancy screening test or lactating or planning to become pregnant in the next 24 months. Female or male patients who were unwilling to use contraceptive methods throughout the study;
9. A history of mental illness;
10. Laboratory tests that meet the following criteria need to be excluded:

(1) Hemoglobin<80g/L; (2) Platelet < 80×109/L; (3) Neutrophil <1.0×109/L; (4) Aspartate aminotransferase (AST) or amino aminotransferase (ALT) > 2.5× upper limit of normal except in relation to the primary disease; 11. Very high-risk patients: presenting with life-threatening nephrotic syndrome, or unexplained rapid deterioration of renal function 12. Any patient judged by the investigator to be unsuitable for inclusion in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-03-29 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The complete response rate at 12 months; | 12 months
  The complete response rate at 12 months;

SECONDARY OUTCOMES:
Response rates at 6, 12, 18 and 24 months (including the proportion of participants with complete response and partial response); | 24 months
  Response rates at 6, 12, 18 and 24 months (including the proportion of participants with complete response and partial response);
Median remission time; | 24 months
  Median remission time;
Proportion of patients without recurrence at 12, 18 and 24 months; | 24 months
  Proportion of patients without recurrence at 12, 18 and 24 months;
Median non-recurrence time; | 24 months
  Median non-recurrence time;
Cumulative dose of glucocorticoids; | 24 months
  Cumulative dose of glucocorticoids;
CD19+ cell count, anti-PLA2R antibody expression level; | 24 months
  CD19+ cell count, anti-PLA2R antibody expression level;
Renal function index: eGFR; | 24 months
  Renal function index: eGFR;
Incidence of adverse events; | 24 months
  Incidence of adverse events;

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Chen, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai Q, Hendricks AR. Membranous nephropathy: A ten-year journey of discoveries. Semin Diagn Pathol. 2020 May;37(3):116-120. doi: 10.1053/j.semdp.2020.01.001. Epub 2020 Jan 29. PMID 32061439
- [Background] Pathological features and diagnosis of membranous nephropathy
- [Background] Dahan K. [Membranous nephropathy: Diagnosis, new insights in pathophysiology, and therapeutic approach]. Rev Med Interne. 2016 Oct;37(10):674-679. doi: 10.1016/j.revmed.2016.02.003. Epub 2016 May 25. French. PMID 27236434
- [Background] Beck LH Jr, Bonegio RG, Lambeau G, Beck DM, Powell DW, Cummins TD, Klein JB, Salant DJ. M-type phospholipase A2 receptor as target antigen in idiopathic membranous nephropathy. N Engl J Med. 2009 Jul 2;361(1):11-21. doi: 10.1056/NEJMoa0810457. PMID 19571279
- [Background] Ruggenenti P, Debiec H, Ruggiero B, Chianca A, Pelle T, Gaspari F, Suardi F, Gagliardini E, Orisio S, Benigni A, Ronco P, Remuzzi G. Anti-Phospholipase A2 Receptor Antibody Titer Predicts Post-Rituximab Outcome of Membranous Nephropathy. J Am Soc Nephrol. 2015 Oct;26(10):2545-58. doi: 10.1681/ASN.2014070640. Epub 2015 Mar 24. PMID 25804280
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Glomerular Diseases Work Group. KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases. Kidney Int. 2021 Oct;100(4S):S1-S276. doi: 10.1016/j.kint.2021.05.021. No abstract available. PMID 34556256
- [Background] Expert consensus on the use of rituximab in glomerulonephritis
- [Background] Expert Group on Biologics Treatment of Immune Glomerular Diseases. Chinese Expert Consensus on Biologics for the Treatment of Immune Glomerular Diseases.
- [Background] Nephrology Expert Panel of the Peking University Health Science Center. [Expert consensus on the application of rituximab in the treatment of membranous nephropathy]. Zhonghua Nei Ke Za Zhi. 2022 Mar 1;61(3):282-290. doi: 10.3760/cma.j.cn112138-20210927-00660. Chinese. PMID 35263969
- [Background] Fervenza FC, Appel GB, Barbour SJ, Rovin BH, Lafayette RA, Aslam N, Jefferson JA, Gipson PE, Rizk DV, Sedor JR, Simon JF, McCarthy ET, Brenchley P, Sethi S, Avila-Casado C, Beanlands H, Lieske JC, Philibert D, Li T, Thomas LF, Green DF, Juncos LA, Beara-Lasic L, Blumenthal SS, Sussman AN, Erickson SB, Hladunewich M, Canetta PA, Hebert LA, Leung N, Radhakrishnan J, Reich HN, Parikh SV, Gipson DS, Lee DK, da Costa BR, Juni P, Cattran DC; MENTOR Investigators. Rituximab or Cyclosporine in the Treatment of Membranous Nephropathy. N Engl J Med. 2019 Jul 4;381(1):36-46. doi: 10.1056/NEJMoa1814427. PMID 31269364
- [Background] Scolari F, Delbarba E, Santoro D, Gesualdo L, Pani A, Dallera N, Mani LY, Santostefano M, Feriozzi S, Quaglia M, Boscutti G, Ferrantelli A, Marcantoni C, Passerini P, Magistroni R, Alberici F, Ghiggeri GM, Ponticelli C, Ravani P; RI-CYCLO Investigators. Rituximab or Cyclophosphamide in the Treatment of Membranous Nephropathy: The RI-CYCLO Randomized Trial. J Am Soc Nephrol. 2021 Apr;32(4):972-982. doi: 10.1681/ASN.2020071091. Epub 2021 Mar 1. PMID 33649098
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Background] Rovin BH, Furie R, Latinis K, Looney RJ, Fervenza FC, Sanchez-Guerrero J, Maciuca R, Zhang D, Garg JP, Brunetta P, Appel G; LUNAR Investigator Group. Efficacy and safety of rituximab in patients with active proliferative lupus nephritis: the Lupus Nephritis Assessment with Rituximab study. Arthritis Rheum. 2012 Apr;64(4):1215-26. doi: 10.1002/art.34359. Epub 2012 Jan 9. PMID 22231479